CLINICAL TRIAL: NCT02191176
Title: A Phase I Multiple Dose Trial to Investigate Safety With Special Emphasis on ECG Effects and Tolerability After Oral Doses of 30 mg q.i.d. and 90 mg q.i.d. Dextromethorphan Hydrobromide Monohydrate (2 mg/mL Syrup) in Healthy Male and Female Subjects for 2 Days Followed by a Morning Dose (Extensive Metabolisers of CYP 2D6) and for 10 Days Followed by a Morning Dose (Poor Metabolisers of CYP 2D6) (Randomised, Double-blind, Placebo-controlled Groups)
Brief Title: Study to Investigate Safety With Special Emphasis on ECG Effects and Tolerability After Oral Doses of Dextromethorphan Hydrobromide Monohydrate in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1134.3
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (3):
- Dextromethorphan syrup - low dose (Experimental)
  Interventions: Drug: Dextromethorphan syrup - low dose
- Dextromethorphan syrup - high dose (Experimental)
  Interventions: Drug: Dextromethorphan syrup - high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dextromethorphan syrup - low dose
  Arms: Dextromethorphan syrup - low dose
Drug: Dextromethorphan syrup - high dose
  Arms: Dextromethorphan syrup - high dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of the current study is to investigate the safety with special emphasis on ECG effects, and tolerability of dextromethorphan hydrobromide monohydrate (2mg/mL syrup) in healthy male and female subjects following oral administration of 30 mg q.i.d. and 90 mg q.i.d. for 2 days followed by a single morning dose (extensive metabolisers of CYP 2D6) and for 10 days followed by a single morning dose (poor metabolisers of CYP 2D6).

Additionally pharmacokinetic properties of dextromethorphan and its main metabolites dextrorphan, 3-hydroxymorphinan, and 3-methoxymorphinan will be investigated

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, oral body temperature, vital signs (blood pressure, pulse rate), 12-lead Electrocardiogram (ECG), clinical laboratory tests
* Age ≥18 and Age ≤55 years
* BMI ≥18.5 and BMI ≤30 kg/m2 (Body Mass Index)
* Extensive or poor metabolisers for CYP 2D6 based on the results of a genotyping test
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within one month prior to first administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to first administration or during the trial)
* Excessive physical activities (within one week prior to first administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QTc interval of >450 ms;
* A history of additional risk factors for Torsades de points (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

Exclusion criteria specific for this study:

* Use of drugs that inhibit or induce cytochrome P 450 enzymes, especially CYP2D6, within 30 days prior to first administration of the study medication or during the trial

For female subjects:

* Pregnancy or planning to become pregnant within 2 months of study completion
* Positive pregnancy test
* No adequate contraception in woman of child bearing potential during the study, i.e., sterilisation, intrauterine device, injectables, oral contraceptive combined with a barrier method of contraception
* Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal findings in physical examination | up to day 20
Number of patients with clinically significant changes in vital signs (blood pressure and pulse rate) | up to day 20
Number of patients with clinically significant changes in 12-lead ECG (electrocardiogram) including QT interval and heart rate corrected QTcN, QTcF (Fridericia) and QTcB (Bazett) | up to day 20
Number of patients with abnormal changes in laboratory parameters | up to day 20
Assessment of tolerability by investigator on a 4-point scale | day 20 (end of trial examination)
Number of patients with adverse events | up to 48 days

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) after the first dose | within 5 hours after first drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) after the first dose | within 5 hours after first drug administration
AUCt1-t2 (area under the concentration-time curve of the analyte in plasma from the time interval t1 to t2) after the first dose | within 5 hours after first drug administration
AUC0-5 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 5 hours after administration) after the first dose | within 5 hours after first drug administration
Cmax,N (maximum measured concentration of the analyte in plasma following the Nth dose) after the last dose | up to day 13
tmax,N (time from last dosing to the maximum concentration of the analyte in plasma following the Nth dose) after the last dose | up to day 13
AUCt1-t2,N (area under the concentration-time curve of the analyte in plasma from the time interval t1 to t2 following the Nth dose) after the last dose | up to day 13
AUC0-5,N (area under the concentration-time curve of the analyte in plasma over the time interval 0 to 5 hours following the Nth dose) after last dose | up to day 13
λz,N (terminal rate constant in plasma following the Nth dose) after the last dose | up to day 13
t1/2,N (terminal half-life of the analyte in plasma following the Nth dose) after the last dose | up to day 13
MRTpo,N (mean residence time of the analyte in the body after oral administration of the Nth dose) after the last dose | up to day 13
Cmax (maximum observed concentration of the analyte in plasma) after the second dose | Day 1
tmax (Time to Cmax of the analyte in plasma) after the second dose | Day 1